CLINICAL TRIAL: NCT00235729
Title: CSP #1024 - A Phase III, Randomized, Multi-Center, Double Blind, Placebo-Controlled Study of Safety and Efficacy of Lofexidine for Relief of Symptoms in Subjects Undergoing Inpatient Opiate Detoxification.
Brief Title: Lofexidine for Inpatient Opiate Detox
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); USWM, LLC (dba US WorldMeds) (Industry)
Responsible Party: Gorodetzky, Charles - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1024; USWM-001
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Opiate Addiction
Keywords: Opiate addiction; Opiate dependence; Withdrawal symptoms
MeSH Terms: conditions — Opioid-Related Disorders; Substance Withdrawal Syndrome | interventions — lofexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Lofexidine 0.8 mg QID
  Interventions: Drug: Lofexidine
- 2 (Placebo Comparator): Placebo QID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lofexidine — Lofexidine is an alpha2-adrenergic-agonist with mild to moderate antihypertensive actions. It is mainly used in the alleviation of opioid withdrawal signs and symptoms.
  Arms: 1
Drug: Placebo — Placebo is an exact match of lofexidine, less the active ingredient.
  Arms: 2

SUMMARY:
The main objective of this study is to investigate the effectiveness of lofexidine in reducing withdrawal symptoms among subjects undergoing opiate detoxification. Currently, lofexidine is the most commonly used non-opiate medication for detoxification from opiates in the United Kingdom (UK). There is no non-opiate medication approved by the Food and Drug Administration (FDA) for the same indication in the United States (US). The only medications currently approved by the FDA for opiate detoxification are methadone and buprenorphine. These medications, however, have the potential to be abused. Lofexidine, on the other hand, offers a unique advantage for opiate detoxification because it is not addicting, is easy to use, and has a favorable safety profile.

DETAILED DESCRIPTION:
Primary Objective: The primary objective of this study is to investigate the efficacy of lofexidine hydrochloride, an alpha-2-adrenergic agonist, in reducing withdrawal symptoms in subjects undergoing opioid detoxification as assessed by 1)Day 3 SOWS-Gossop score during treatment phase, and 2)Time to dropout during treatment phase.

Secondary Objectives: Secondary objectives include determining Lofexidine's: 1) Efficacy in the reduction in withdrawal symptoms in subjects undergoing opioid detoxification (assessed by longitudinal changes in SOWS-Gossop, OOWS-Handelsman, VAS-E and MGCI (subject and rater); 2)Efficacy in the reduction in the need of any concomitant medication to alleviate opiate withdrawal symptoms: 3) Efficacy in increasing the number of completers during the treatment phase; and 4) Safety in the study population.

Study Design: This is a randomized, multi-center, double blind, placebo-controlled, parallel-group study. There are 3 major phases of the study. During Phase I (Screening) screening assessments will be performed; during Phase II (Days 1-5), subjects will be admitted to an inpatient unit and randomized to receive either lofexidine (0.8 mg QID) or placebo QID after the baseline assessments are performed prior to randomization on Day 1; and during Phase III (Days 6-8), all subjects will receive placebo QID on Days 6-7, and then be discharged on Day 8 following the post-treatment assessments. An adaptive randomization procedure will be used to randomly allocate subjects in one of the two treatment groups - lofexidine or placebo.

Study Population: 264 subjects with Diagnostic and Statistical Manual for Mental Disorders Fourth Edition (DSM-IV) criteria for current dependence on any opioid with a half-life similar to heroin or morphine determined by structured clinical interview (SCID) will be randomized in one of the treatment groups (132 subjects per group). Subjects at least 18 years-of-age with positive urine toxicology screen for opiates and negative for methadone, LAM/LAAM, or buprenorphine during screening, with the ability to understand and provide written informed consent that meet all the inclusion criteria and do not meet any of the exclusion criteria may be randomized into the study.

Treatments: On Day 1, subjects are randomized to either lofexidine or placebo and receive lofexidine (0.8 mg [4 x 0.2 mg lofexidine tablets] QID) or placebo (4 matching placebo tablets QID). Lofexidine or placebo will be administered orally within 15 minutes before or after 0800, 1300, 1800 and 2300 hours on Days 1-5. On Days 6 and 7, all subjects will receive placebo using the same dosing schedule as above.

Efficacy Assessments: The primary efficacy outcome measures will be the Short Opiate Withdrawal Scale (SOWS-Gossop) scores (range = 0-30) on Day 3 of the treatment phase defined as Days 1-5, and the number of days representing the duration of stay in the treatment program after randomization. SOWS-Gossop will be administered once during Baseline on Day 1 prior to randomization and after 3.5 hours after the first dose on Days 1 - 7. Secondary outcome measures evaluating the treatment effects on opioid withdrawal symptoms include, the proportion of subjects requiring any concomitant medication to alleviate opiate withdrawal symptoms and the proportion of subjects who are completers. In addition, the composite longitudinal scores of the SOWS-Gossop, Objective Opiate Withdrawal Scale (OOWS-Handelsman), Modified Global Clinical Impression Scale (Subject and Rater), and Visual Analog Scale - Efficacy (VAS-E) will also be used to assess the treatment efficacy to reduce the withdrawal symptoms. OOWS-Handelsman, MGCI (Subject and Rater), and VAS-E will be administered once during Baseline on Day 1 prior to randomization and 3.5 hours after the first dose on Days 1-7.

Safety Assessments: After signing the informed consent and completing the consent quiz, the subject will complete Screening assessments to determine eligibility for study enrollment. A complete physical examination will be performed on the first day of screening. A repeat physical exam will be performed at 3-4 hours after randomization on Day 1, and prior to discharge on Day 8 or at early termination. A 12-lead ECG will be conducted on the first day of screening and immediately prior to admission. Four hours after receiving the first dose of study medication on Days 1-7, a 12-lead ECG will also be conducted. A 12-lead ECG will be done prior to discharge on Day 8 or at early termination. If, in the opinion of the investigator, clinically significant changes are noted on the ECG, these measurements should be performed more frequently. Additionally, the next scheduled dose of study medication may be withheld at the discretion of the investigator, or the subject may be discontinued from the study. Subjects will be awakened and weighed each morning prior to breakfast. Vital signs (systolic and diastolic blood pressure, heart rate, respiration rate, and body temperature) are to be measured 3 hours after each dose of study medication at 0800, 1300, and 1800 on Days 1-7, and prior to discharge on Day 8. For the orthostatic blood pressure readings, subjects will remain sitting for 3 minutes prior to a blood pressure reading, and then stand for 1 minute prior to a second blood pressure reading. Clinical lab tests will be done during Screening, on Day 7 or early termination, and as needed at the physician?s discretion. The urine sample collected on the first day of Screening will be divided into two aliquots. One sample will go to the local lab for confirmatory drug testing. The other sample will be used for immediate "dip-stick" analysis of pregnancy (for the female patients only). A second "dip-stick" pregnancy test will be done during Baseline, prior to randomization. Adverse events and concomitant medication use will be assessed every day during the study (Days 1-8).

Subjects who demonstrate symptoms of withdrawal will be treated with a standard of care using the concomitant medications listed in Section 13.11. At subject?s request, and at any time, subject can be discontinued from the study without prejudice, and will be medically stabilized; subject will then be referred, at subject's expense, for further treatment.

Analysis: The primary outcome measures and each of the secondary outcome measures will be analyzed using appropriate statistical methods for the intent-to-treat, the evaluable and for the completer groups. The Intent-to-Treat (ITT) group is defined as the subjects who are randomized to treatment. The evaluable group is defined as subjects in the ITT group who receive at least one dose of study medication and complete the post-medication SOWS on Day 1. The completer group will consist of all patients in the ITT group who meet the following criteria: receive at least one dose of study drug on Day 5, and complete the SOWS-Gossop assessment on Day 5.

It is hypothesized that lofexidine treatment, compared to placebo, will be associated with a significant reduction in opiate withdrawal symptoms. All statistical tests will be two-sided at 5% Type-I error rate. Confidence intervals will be two-sided with a 95% confidence coefficient.

Summaries of the characteristics of the subject population in both treatment groups at baseline will be prepared for the modified intent-to-treat group and the completer group. A summary will be prepared to show dropouts/retention over time in each group and for subpopulations. All adverse events will be reported quarterly indicating the counts of unique adverse events by body system and preferred term (MedDRA coded) as experienced by study subjects in both the groups. Laboratory data, physical examinations, and vital signs will be reported in tabular form.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must:

1. Be at least 18 years of age.
2. Have current dependence, according to SCID criteria, on any opioid with a half-life similar to heroin or morphine, including Vicodin, Lortab, or Lorcet, Percocet, Percodan, Tylox, or Hydrocodone (by any route of administration), or oxycodone (oxycodone and oxycodone time-released formulation when crushed and snorted, injected or swallowed after chewing).
3. Be seeking treatment for opiate dependence.
4. Have a score greater than or equal to 2 on the Objective Opiate Withdrawal Scale-Handelsman (OOWS) immediately prior to admission.
5. Have reported use of heroin, morphine, or any opioid with a half-life similar to heroin or morphine, for at least 21 of the past 30 days.
6. Have urine toxicology screen positive for opiates and negative for methadone or buprenorphine.
7. If female and of child bearing potential, agree to use of one of the following methods of birth control:

   1. oral contraceptives
   2. patch
   3. barrier (diaphragm, sponge or condom) plus spermicidal preparations
   4. intrauterine contraceptive system
   5. levonorgestrel implant
   6. medroxyprogesterone acetate contraceptive injection
   7. complete abstinence from sexual intercourse
   8. hormonal vaginal contraceptive ring
   9. surgical sterilization or partner sterile (must have documented proof)
8. Have completed the ASI during screening and all other assessments (SOWS-Gossop OOWS, and MCGI) during the baseline period.
9. Be able to verbalize understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures and pass the study consent quiz with 100% accuracy (if necessary, quiz may be administered more than one time).

Exclusion Criteria:

Potential subjects must not:

1. Be female subjects who are pregnant or lactating.
2. Have self-reported use of methadone or buprenorphine in the past 14 days.
3. Have serious medical illnesses including, but not limited to:

   1. Seizures, or those who have received anticonvulsant therapy during the past 5 years.
   2. Pancreatic disease such as insulin-dependent diabetes.
   3. Liver disease requiring medication or medical treatment, and/or aspartate or alanine aminotransferase levels greater than 5 times the upper limit of normal.
   4. Gastrointestinal or renal disease, which would significantly impair absorption, metabolism or excretion of study drug, or would require medication or medical treatment.
4. Have a psychiatric disorder, as assessed by the SCID, including but not limited to dementia or any disorder that, in the opinion of the study physician requires ongoing treatment that would make study participation unsafe or which would make treatment compliance difficult.
5. Have self-reported AIDS.
6. Have an abnormal cardiovascular exam prior to randomization, including any of the following:

   1. Clinically significant abnormal ECG (e.g., second or third degree heart block, uncontrolled arrhythmia, or QTc interval > 450 msec for males, and > 470 msec for females).
   2. Heart rate less than 45 bpm or symptomatic bradycardia.
   3. Systolic blood pressure < 90 mm Hg or symptomatic hypotension (diastolic blood pressure < 60 mm Hg).
   4. Blood pressure > 160/100 mm Hg.
   5. Prior history of myocardial infarction.
7. Have clinically significant abnormal laboratory values.
8. Require any of the following medications currently or within the past 4 weeks: psychotropics (including sedatives/hypnotics, antidepressants, neuroleptics), prescription analgesics (excluding those listed in inclusion criteria #2 above), anticonvulsants, antihypertensives, antiarrhythmics, antiretroviral, and cholesterol lowering medications. Nicotine replacement therapy (patch, inhaler, gum, or nasal spray) for nicotine-dependent subjects are allowed.
9. Have current dependence (by SCID criteria) on

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2006-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
SOWS-Gossop score on Day 3 during the treatment phase & time-to-dropout for the subjects in the two treatment groups. during the treatment phase. | Day 3 of treatment phase for the SOWs score. Time to dropout will be measured as the number of 6-hour time quadrants until a subject withdraws or completes the treatment phase of the study

CONTACTS AND LOCATIONS:
Overall Officials: Charles W. Gorodetzky, Study Chair — VA Maryland Health Care System, Baltimore
Locations (16):
- United States (16):
  - CNS, Cerritos, Cerritos, California
  - CNS Psychiatric Institute of Washington, Washington D.C., District of Columbia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Alexian Center for Psychiatric Research, Hoffman Estates, Illinois
  - University of Kentucky, Lexington, Kentucky
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - Wayne State University School of Medicine, Detroit, Michigan
  - Richmond Medical Center, Staten Island, New York
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - VA Medical Center, Providence, Providence, Rhode Island
  - Psychiatric Hospital at Vanderbilt, Nashville, Tennessee
  - Research Across America, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington
  - Aurora Psychiatric Hospital, Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Alam D, Tirado C, Pirner M, Clinch T. Efficacy of lofexidine for mitigating opioid withdrawal symptoms: results from two randomized, placebo-controlled trials. J Drug Assess. 2020 Jan 8;9(1):13-19. doi: 10.1080/21556660.2019.1704416. eCollection 2020. PMID 32002194